CLINICAL TRIAL: NCT02098265
Title: A Closed Loop Neural Activity Triggered Stroke Rehabilitation Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0469; A539300 (Other: UW Madison); SMPH/RADIOLOGY (Other: UW Madison); 15GRNT25780033 (Other Grant/Funding Number: American Heart Association); Protocol Version 2/1/22 (Other: UW Madison)
Record Dates: First submitted 2014-03-06; First posted 2014-03-27 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: aneurysm; transient ischemic attack
MeSH Terms: conditions — Stroke; Aneurysm; Ischemic Attack, Transient | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Experimental Group - Immediate BCI Therapy (Experimental): EEG - BCI training (closed loop)
  Interventions: Behavioral: Behavioral Assessments; Other: Magnetic Resonance Imaging; Other: EEG; Device: BCI-FES
- Experimental Group - Delayed BCI Therapy (Experimental): Scanned and tested 4 times over a 10-week period before EEG-BCI training
  Interventions: Behavioral: Behavioral Assessments; Other: Magnetic Resonance Imaging; Other: EEG; Other: Delay; Device: BCI-FES
- Experimental Group - RecoveriX (Experimental): Recruited from participants who have completed the study intervention
  Interventions: Other: RecoveriX
- Control Group 1 (Active Comparator): 48 stroke patients, 48 participants with risk factors for stroke, 48 healthy controls receiving 4-6 training sessions on the EEG-BCI, pre- and post- behavioral testing, and MRI
  Interventions: Behavioral: Behavioral Assessments; Other: Magnetic Resonance Imaging; Other: EEG; Device: BCI-FES
- Control Group 2 (Active Comparator): 24 Stroke Patients with UE impairment receiving standard FES only therapy
  Interventions: Device: Functional Electric Stimulation (FES)

INTERVENTIONS:
Device: Functional Electric Stimulation (FES) — FES uses low energy electrical pulses to artificially generate body movements in individuals with muscle paralysis. FES can be used to generate muscle contraction in otherwise paralyzed limbs to restore function.
  Arms: Control Group 2
Behavioral: Behavioral Assessments — These assessments will include measures of upper extremity motor assessments, standard stroke scales, and measures of activities of daily living.
  Arms: Control Group 1; Experimental Group - Delayed BCI Therapy; Experimental Group - Immediate BCI Therapy
Other: Magnetic Resonance Imaging — A functional magnetic resonance image will be collected.
  Arms: Control Group 1; Experimental Group - Delayed BCI Therapy; Experimental Group - Immediate BCI Therapy
Other: EEG — EEG electrodes will be attached to the participant's scalp using a standard, commercially available electrode cap. Proper electrode placement is made according to the international 10-20 system, ensuring complete electrode coverage over sensorimotor cortex.
  Other Names: Electroencephalography
  Arms: Control Group 1; Experimental Group - Delayed BCI Therapy; Experimental Group - Immediate BCI Therapy
Other: RecoveriX — RecoveriX is a brain driven rehabilitation system for stroke patients that pairs mental activities with motor functions.
  Arms: Experimental Group - RecoveriX
Other: Delay — 10 week delay before intervention
  Arms: Experimental Group - Delayed BCI Therapy
Device: BCI-FES
  Arms: Control Group 1; Experimental Group - Delayed BCI Therapy; Experimental Group - Immediate BCI Therapy

SUMMARY:
The purpose of this research is to determine if two non-invasive brain stimulation techniques, muscle stimulation of the arm and neuro-stimulation through the tongue, can increase the extent of stroke recovery.

DETAILED DESCRIPTION:
The aim of this study is to determine if functional muscle stimulation, in addition to non-invasive neurostimulation through the tongue (TDU), directed by electroencephalogram (EEG) output, can increase the extent of stroke recovery on behavioral measures and induce brain plasticity as measured by functional magnetic resonance imaging (fMRI).

Adult stroke patients with upper extremity motor impairments (henceforth "experimental group"), healthy controls, and participants with risk factors for stroke, without upper extremity impairment (allowing them to serve as controls for patients with upper extremity impairments (henceforth "control group")), will be recruited in this study. Half of the participants in the experimental group will be randomly assigned to the EEG-BCI (brain-computer interface) training ("closed-loop") group and will receive training on the BCI task along with muscle and tongue stimulation. The other half of the participants in the experimental group receiving traditional rehab will not receive any kind of FES or tongue stimulation for the first 8-10 weeks of study period and then will start receiving BCI-FES-tongue stimulation rehab therapy.

All participants without UE impairment in Control group 1 will receive 4-6 (minimum 4, up to a maximum of 6) sessions of training on the BCI system and pre- and post MRI and 2 behavioral testing sessions.

Addition of a Control group 2 is consistent with the AHA grants - Twenty four ischemic stroke patients with moderate upper extremity (dominant right hand affected) impairment (score of 1 or 2 on the motor sub-component of the NIH stroke scale (NIHSS) and ARAT score 20-45); no upper extremity injury or conditions that limited use prior to the stroke; and pre-stroke independence with a Modified Rankin Score of 0 or 1), will be recruited in this arm. All participants in this group will receive MR sessions and behavioral testing similar to the Experimental group.

Addition of an Experimental group receiving EEG-BCI-bilateral FES intervention using the recoveriX system: recoveriX is a brain driven rehabilitation system for stroke patients that pairs mental activities with motor functions. Through the EEG-based recoveriX BCI system, the brain receives visual and tactile feedback in real-time, making rehabilitation more effective. A stroke patient imagines a hand movement while receiving visual feedback through a virtual avatar, and tactile feedback through electrical muscle stimulation paired to the patient's imagined movement, with the aim that these patients might regain the volitional ability to grasp following therapy. Unlike the current EEG-BCI-FES intervention that involves stimulation of only the impaired arm, with recoveriX, both arms are simultaneously stimulated during the course of the intervention.

Specific Aims

To determine if functional muscle stimulation of the arms, in addition to non-invasive neurostimulation through the tongue (TDU), directed by electroencephalogram (EEG) output, can increase the extent of stroke recovery as measured by behavioral measures and induce brain plasticity as measured by functional magnetic resonance imaging (fMRI).

Primary objective

* To examine the effect of EEG guided functional muscle stimulation on improvement in upper extremity function

Secondary objective

* To examine plasticity changes as measured by EEG/fMRI measures before and after EEG guided functional muscle stimulation.

ELIGIBILITY:
Inclusion Criteria (Experimental Group):

* Stroke patients with persistent upper extremity (UE) deficits

Inclusion Criteria (Control Group 1)

* Stroke patients without UE impairments
* Participants with risk factors for stroke
* healthy controls

  * No known neurologic, psychiatric or developmental disability

Inclusion Criteria (Control Group 2)

* Stroke patients with persistent upper extremity (UE) deficits
* Moderate upper extremity (dominant right hand affected) impairment (score of 1 or 2 on the motor sub-component of the NIH stroke scale (NIHSS) and ARAT score 20-45)
* No upper extremity injury or conditions that limited use prior to the stroke
* Pre-stroke independence with a Modified Rankin Score of 0 or 1, for the standard FES only intervention.

Exclusion Criteria (for all participants):

* Allergic to electrode gel, surgical tape and metals
* Participants under treatment for infectious diseases or having apparent oral lesions or inflammation will be excluded from the study
* Women who are pregnant or may become pregnant during the course of the study will be excluded
* Participants with contraindications for MRI will be offered the opportunity to participate in the interventions study only (e.g. EEG-BCI-FES and behavioral testing)

Exclusion Criteria (for healthy controls)

* Contraindications for MRI
* Allergic to electrode gel, surgical tape, and metals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2010-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test Scores | 4 months
  The Action Research Arm Test (ARAT) is designed for evaluation of upper extremity function. This test consists of sections for Grasp, Grip, Pinch and Gross Movements and comprise a total of 19 tests. Each test is scored 0-3 where 0 is 'no movement' and 3 is 'the movement is performed normally'. Each section is scored separately and the scores added for a total possible range of scores from 0-57 where the higher the score, the complete and efficient the movement. ARAT will be assessed at baseline and end of study (approximately 4 months)

SECONDARY OUTCOMES:
Change in Electroencephalogram (EEG) Response Strength | 4 months
  The change in the strength of the EEG response before and after functional stimulation during left arm imagery with respect to right arm imagery.
Signal change in functional MRI | 4 months
  To compare the percent signal change in the functional MRI activations before and after functional stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Prabhakaran, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Young BM, Stamm JM, Song J, Remsik AB, Nair VA, Tyler ME, Edwards DF, Caldera K, Sattin JA, Williams JC, Prabhakaran V. Brain-Computer Interface Training after Stroke Affects Patterns of Brain-Behavior Relationships in Corticospinal Motor Fibers. Front Hum Neurosci. 2016 Sep 16;10:457. doi: 10.3389/fnhum.2016.00457. eCollection 2016. PMID 27695404
- [Result] Young BM, Nigogosyan Z, Walton LM, Remsik A, Song J, Nair VA, Tyler ME, Edwards DF, Caldera K, Sattin JA, Williams JC, Prabhakaran V. Dose-response relationships using brain-computer interface technology impact stroke rehabilitation. Front Hum Neurosci. 2015 Jun 23;9:361. doi: 10.3389/fnhum.2015.00361. eCollection 2015. PMID 26157378
- [Result] Song J, Nair VA, Young BM, Walton LM, Nigogosyan Z, Remsik A, Tyler ME, Farrar-Edwards D, Caldera KE, Sattin JA, Williams JC, Prabhakaran V. DTI measures track and predict motor function outcomes in stroke rehabilitation utilizing BCI technology. Front Hum Neurosci. 2015 Apr 27;9:195. doi: 10.3389/fnhum.2015.00195. eCollection 2015. PMID 25964753
- [Result] Song J, Young BM, Nigogosyan Z, Walton LM, Nair VA, Grogan SW, Tyler ME, Farrar-Edwards D, Caldera KE, Sattin JA, Williams JC, Prabhakaran V. Characterizing relationships of DTI, fMRI, and motor recovery in stroke rehabilitation utilizing brain-computer interface technology. Front Neuroeng. 2014 Jul 29;7:31. doi: 10.3389/fneng.2014.00031. eCollection 2014. PMID 25120466
- [Result] Young BM, Nigogosyan Z, Nair VA, Walton LM, Song J, Tyler ME, Edwards DF, Caldera K, Sattin JA, Williams JC, Prabhakaran V. Case report: post-stroke interventional BCI rehabilitation in an individual with preexisting sensorineural disability. Front Neuroeng. 2014 Jun 24;7:18. doi: 10.3389/fneng.2014.00018. eCollection 2014. PMID 25009491
- [Derived] Remsik AB, Williams L Jr, Gjini K, Dodd K, Thoma J, Jacobson T, Walczak M, McMillan M, Rajan S, Young BM, Nigogosyan Z, Advani H, Mohanty R, Tellapragada N, Allen J, Mazrooyisebdani M, Walton LM, van Kan PLE, Kang TJ, Sattin JA, Nair VA, Edwards DF, Williams JC, Prabhakaran V. Ipsilesional Mu Rhythm Desynchronization and Changes in Motor Behavior Following Post Stroke BCI Intervention for Motor Rehabilitation. Front Neurosci. 2019 Mar 6;13:53. doi: 10.3389/fnins.2019.00053. eCollection 2019. PMID 30899211
- [Derived] Remsik AB, Dodd K, Williams L Jr, Thoma J, Jacobson T, Allen JD, Advani H, Mohanty R, McMillan M, Rajan S, Walczak M, Young BM, Nigogosyan Z, Rivera CA, Mazrooyisebdani M, Tellapragada N, Walton LM, Gjini K, van Kan PLE, Kang TJ, Sattin JA, Nair VA, Edwards DF, Williams JC, Prabhakaran V. Behavioral Outcomes Following Brain-Computer Interface Intervention for Upper Extremity Rehabilitation in Stroke: A Randomized Controlled Trial. Front Neurosci. 2018 Nov 8;12:752. doi: 10.3389/fnins.2018.00752. eCollection 2018. PMID 30467461
- See also: Publication resulting from this work. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5025476/
- See also: Publication resulting from this work. — https://www.ncbi.nlm.nih.gov/pubmed/26157378
- See also: Publication resulting from this work. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4410488/
- See also: Publication resulting from this work. — https://www.ncbi.nlm.nih.gov/pubmed/25120466
- See also: Publication resulting from this work. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4067954/